CLINICAL TRIAL: NCT02626273
Title: ADIposity and Bone Metabolism: Effects of eXercise-induced Weight Loss in Obese Adolescents
Acronym: ADIBOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other); Australian Catholic University (Other); Tza Nou Medical House for children and adolescents, 230, rue Vercingétorix - B.P. 77 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-0249; 2015-A01024-45 (Registry Identifier: 2015-A01024-45)
Record Dates: First submitted 2015-11-03; First posted 2015-12-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: obesity; adolescents; physical activity; adipocytes; osteocytes; weight loss; bone; fat
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss; Platelet Glycoprotein IV Deficiency

ARMS (2):
- intervention group (Experimental): an intervention group who will undergo the management program combining physical activity and restrictive diet at Tza Nou Medical House for 10 months
  Interventions: Radiation: weight loss
- a control group (Other): a control group who will not undergo any intervention
  Interventions: Radiation: weight loss

INTERVENTIONS:
Radiation: weight loss

SUMMARY:
The present protocol is mainly involved in the understanding of the local interaction between the released products by fat tissue and hormones production of bone tissue. These complex interactions between adipocyte and osteocyte activities could explain the mechanisms of the body responses to the strategies of weight loss that include diet and/or physical activity program, as well as the side effects encountered by these interventions.

Adolescence is a period of development characterized by many metabolic and somatic changes that may influence weight. Weights bearing physical activities are a key factor allowing body composition changes (i.e. fat and bone tissue). The difficulties of managing weight and the onset of overweight and obesity during this very important growth spurt lead to various hormonal dysregulation. The specific mechanisms of the evolution and interactions between these two parameters (fat and bone tissue) are not yet elucidated; therefore our aim is to analyze the possible connections between fat tissue and the quality of the skeleton in order to reduce related risks of the consequence of weight loss in obese individuals.

DETAILED DESCRIPTION:
The complex consequences of childhood obesity represent major concerns in most developed countries, largely contributing to metabolic complications with costly repercussions for the burden of disease. The burden is exemplified by high prevalence rates of overweight or obesity.

The ADIBOX protocol was designed to provide a better understanding of the bone-adipocyte cross-talk in adolescents with obesity and the effects of physical activity-induced weight loss on this cross-talk.

Obesity effectively leads to hormonal alterations favoring the accumulation of fat mass and loss of bone mass. Advancing the knowledge of the complex interactions between adipocyte and osteocyte activities may contribute to the mechanistic understanding of the body's responses to weight loss during adolescence and prevent cardiovascular risk. Indeed, the adipose-bone tissue cross-talk has been recently linked with cardiovascular diseases. Similarly as adipose tissue, released-products from bone tissue may act directly or indirectly on cardiovascular risk and diseases.

The ADIBOX study, a 40 weeks longitudinal study (LS) with repeated measures on four occasions (baseline and every fourteen weeks), will allow us to understand the effects of physical activity-induced weight loss on this cross-talk in obese adolescents.

Data will be analyzed using Stata (StataCorp, College Station, USA) and IBM Statistics SPSS version 22 (IBM Corp, 2013, Chicago, IL, USA) and significance will be accepted at a two-sided alpha level of p<0.05. After testing for normal distribution (Shapiro-Wilk test), data will be treated either by parametric or non-parametric analyses according to statistical assumptions.

Student t tests or Mann-Whitney U test will be performed to compare adipose tissue (total, subcutaneous, visceral) variation reported to bone mass variation at lumbar spine between groups at baseline. Pearson (or Spearman when appropriate) correlation coefficient will be used and compared with Fisher test (command corcor Stata) to measure the link between exercise-inducing weight loss on adipose tissue and bone mass variations. Longitudinal data will be treated using a mixed model analyses in order to treat fixed effects group, time and group x time interaction taking into account between and within participant variability.

ELIGIBILITY:
Inclusion Criteria:

* All adolescent girls will have to be free of any recent history of hospitalization (past two years) or of systemic illness lasting more than two weeks in the past 12 months. .

Exclusion Criteria:

* pregnant girl
* diabetes
* insulin-resistance
* hypo or hyper-thyroid
* consuming alcohol
* smokers

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
change from baseline fat mass measured by Dual energy X-ray Absorptiometry (DXA) | at 10 months.
change from baseline bone mass measured by Dual energy X-ray Absorptiometry (DXA) | at 10 months

SECONDARY OUTCOMES:
Whole body measured by Dual energy X-ray Absorptiometry (DXA) | at 10 months
weight waist | at 10 months.
waist circumference | at 10 months.
lower limb bone lengths | at 10 months.
Physical activity measured with International Physical Activity Questionnaire | at 10 months.
Tanner's stages model for pubertal maturation | at 10 months.
Energy metabolism assessed by cycle-ergometer submaximal aerobic fitness | at 10 months.
bone mineral density measured by Peripheral Quantitative Computed Tomography | at 10 months.
bone mineral status measured by Quantitative Ultra-Sound (QUS) on the non-dominant calcaneus. | at 10 months.
Endocrine assays | at 10 months.
Adolescents' observance to the weight loss lifestyle program | at 10 months
Metabolomics analysis in blood plasma | at 10 months
Ex-vivo mechanistic analysis | at 10 months
left ventricular end diastolic diameter measured by echocardiography | at 10 months
left ventricular end systolic diameter measured by echocardiography | at 10 months
posterior wall thickness measured by echocardiography | at 10 months
interventricular septum thickness measured by echocardiography | at 10 months
left ventricular mass indexed measured by echocardiography | at 10 months
left ventricular ejection fraction measured by echocardiography | at 10 months
valves velocity measured by echocardiography | at 10 months
isovolumic relaxation time measured by echocardiography | at 10 months
strain rate measured by echocardiography | at 10 months
myocardial dyssynchrony measured by echocardiography | at 10 months
carotid-intima-media thickness measured by echography | at 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Chaplais E, Dutheil F, Naughton G, Greene D, Pereira B, Thivel D, Courteix D. Cross-sectional and longitudinal study protocols of the 'ADIposity and BOne metabolism: effects of eXercise-induced weight loss in obese adolescents' (ADIBOX) project. BMJ Open. 2016 Oct 18;6(10):e011407. doi: 10.1136/bmjopen-2016-011407. PMID 27797988